CLINICAL TRIAL: NCT02320851
Title: Tailored Care for Somatoform Vertigo/Dizziness - From Diagnostics to Therapy
Brief Title: Tailored Care for Somatoform Vertigo/Dizziness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Technical University of Munich (Other)
Collaborators: German Center for Vertigo and Balance Disorders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01EO1401
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Somatoform Vertigo/Dizziness
Keywords: Somatoform disorder; Functional vertigo/dizziness; Chronic subjective dizziness
MeSH Terms: conditions — Dizziness; Somatoform Disorders | interventions — Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SVD-tailored Integrative Psychotherapy (IPT) (Experimental): IPT is a short-term psychotherapy aiming to ameliorate both physical and psychosocial distress. It emanates from a multidirectional and dynamic relationship among body, mind, and environment irrespective of causality. In a multi-component approach, other elements are integrated into it, such as cognitive-behavioral and psychodynamic techniques, psychoeducation and body-oriented techniques. The IPT intervention tailored to SVD will be delivered for 16 weeks in a manualised setting with one group session per week (à 90 minutes) and one additional booster session three months after the end of the therapy. The group psychotherapy is on a 6-8:1 basis and will be conducted by a psychotherapist trained on the basis of the manual and under regular clinical supervision.
  Interventions: Behavioral: SVD-tailored Integrative Psychotherapy (IPT)
- Self-help group (SHG) (Active Comparator): The experimental condition will be compared to moderated self-help groups without the implementation of additional therapeutic interventions. Those can be classified as low-level non-placebo control. Treatment will consist of 16 weekly moderated SHG sessions (one weekly session à 90 minutes) and one additional booster-session at three months after the end of the control intervention to be delivered on a 6-8:1 basis by a trained SHG moderator under clinical supervision.
  Interventions: Behavioral: Self-help group (SHG)

INTERVENTIONS:
Behavioral: SVD-tailored Integrative Psychotherapy (IPT) — (see description of corresponding study arm)
  Arms: SVD-tailored Integrative Psychotherapy (IPT)
Behavioral: Self-help group (SHG) — (see description of corresponding study arm)
  Arms: Self-help group (SHG)

SUMMARY:
The purpose of this study is to evaluate the efficacy of a manualised, multimodal group psychotherapy, based on integrative psychotherapy (IPT) and tailored to somatoform vertigo/dizziness (SVD) subgroups of mental disorders, compared to self-help groups (SHGs) in patients with SVD. The investigators hypothesise that patients who received IPT will demonstrate greater improvement concerning their vertigo-related handicap compared to patients from the SHGs. The investigators will also analyse the cost-effectiveness of experimental and control intervention.

DETAILED DESCRIPTION:
Vertigo/dizziness (VD) is one of the most frequent problems in medicine with a one-year prevalence of 23%. Approximately 50% of the complex VD disorders (i.e., VD is the cardinal symptom and persists > 6 months) are not fully explained by an identifiable medical condition and could be labelled as somatoform vertigo/dizziness (SVD), fulfilling the criteria of somatoform disorder according to ICD-10 or DSM-IV, respectively. SVD shows a high comorbidity rate of other mental disorders, such as anxiety/phobic and depressive disorders. The majority of the patients with SVD suffer severe impairments in their daily and working lives and report a poorer quality of life compared to the patients with organic VD. Although preliminary evidence indicates that psychotherapy may be effective in these patients, the therapeutic options in the treatment of SVD remain unsatisfactory.

In this two-armed, single-centre, randomised, controlled, open superiority clinical trial, the long-term efficacy of manualised, multimodal group psychotherapy, based on integrative psychotherapy (IPT) and tailored to SVD subgroups of mental disorders will be investigated in patients with SVD compared to self-help groups (SHGs). IPT describes a differentiated psychotherapeutic approach, which combines different therapeutic techniques, such as interpersonal skills and psychodynamic aspects, self-management and symptom management skills, psychoeducation, and relaxation techniques. Within this study, IPT is tailored to SVD including its common mental comorbidity.

Patients will be recruited via routine care appointments at the German Centre for Vertigo and Balance Disorders, a specialised tertiary care unit at the Klinikum Großhadern (Ludwig-Maximilians-Universitaet, Munich).

Our principal research questions are as follows: Will IPT result in a clinically relevant improvement in vertigo/dizziness-related quality of life? Does this long-term improvement also apply to associated mental symptoms, such as depression, anxiety and somatisation, as well as balance strategies measured by posturography? Is IPT in the long term superior to moderated SVD-SHGs? The investigators hypothesise that the patients who received IPT will demonstrate greater improvement concerning their vertigo-related handicap compared to the patients from the SHGs. The investigators will also analyse the cost-effectiveness of this trial.

ELIGIBILITY:
Inclusion Criteria:

* SVD diagnosis
* Clinically relevant SVD (VHQ sum score > 45)
* Informed consent

Exclusion Criteria:

* Insufficient German language ability
* Insufficient cognitive abilities (Mini Mental State Test (MMST) ≤ 27)
* Severe and chronic comorbid somatic or mental disease (e.g., suicidality, severe depression, drug addiction)
* Current psychotherapeutic treatment
* Living > 50 km away from Munich

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-07 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Vertigo-related quality of life | Improvement at follow-up (12 months after treatment)
  Absolute improvement of vertigo-related quality of life on the Vertigo Handicap Questionnaire (VHQ) at 12 months after the 16-week therapy sessions from VHQ at randomisation/baseline.

SECONDARY OUTCOMES:
Generic quality of life | Improvement at follow-up (12 months after treatment)
  Generic quality of life will be measured using the Quality of Life Questionnaire (EQ-5D).
Severity of vertigo | Improvement at follow-up (12 months after treatment)
  Severity of vertigo will be measured using the Vertigo Symptom Scale (VSS).
Depression | Improvement at follow-up (12 months after treatment)
  Depression will be measured using the Beck Depression Inventory (BDI-II).
Anxiety | Improvement at follow-up (12 months after treatment)
  Anxiety will be measured using the Beck Anxiety Inventory (BAI).
Somatisation | Improvement at follow-up (12 months after treatment)
  Somatisation will be measured using the Patient Health Questionnaire 15 (PHQ-15).
Computerized Static Posturography and Head Impulse Test | Improvement at follow-up (12 months after treatment)
  Both assessments (Computerized Static Posturography and Head Impulse Test) are introduced as state-of-the-art validated objective dimensions that address relevant core elements of the study conditions and allow for the estimation of possible intervention effects independent from the patients' self-reported outcomes.

OTHER OUTCOMES:
Cost-effectiveness | Baseline and follow-up (12 months after treatment)
  Cost-effectiveness will be measured as quality-adjusted life years (QALYs) derived from the EQ-5D at baseline and at 12 months after the 16-week therapy sessions. Costs related to absence from work and health care utilisation will be obtained using a modified German version of the Trimbos/iMTA questionnaire for costs associated with Psychiatric Illness (TiC-P).

CONTACTS AND LOCATIONS:
Overall Officials: Claas Lahmann, PD Dr. med., Principal Investigator — Department of Psychosomatic Medicine and Psychotherapy, Klinikum rechts der Isar, Technische Universitaet, Munich

REFERENCES:
- [Derived] Limburg K, Radziej K, Sattel H, Henningsen P, Dieterich M, Probst T, Dale R, Lahmann C. A Randomized Controlled Trial Evaluating Integrative Psychotherapeutic Group Treatment Compared to Self-Help Groups in Functional Vertigo/Dizziness. J Clin Med. 2021 May 20;10(10):2215. doi: 10.3390/jcm10102215. PMID 34065517
- [Derived] Lahmann C, Henningsen P, Dieterich M, Radziej K, Schmid G. Tailored care for somatoform vertigo/dizziness: study protocol for a randomised controlled trial evaluating integrative group psychotherapy. J Neurol. 2015 Aug;262(8):1867-75. doi: 10.1007/s00415-015-7784-6. Epub 2015 May 23. PMID 26001913